CLINICAL TRIAL: NCT05800197
Title: Neoadjuvant Endocrine Therapy in Breast Cancer. Real Clinical Practice in Russia
Acronym: NEMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Blokhin's Russian Cancer Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: 17.03.2023
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer; Neoadjuvant Endocrine Therapy
Keywords: Breast Cancer; Neoadjuvant Endocrine Therapy; postmenopausal women; premenopausal women
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Anastrozole; Letrozole; Goserelin; Triptorelin Pamoate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- premenopausal women: premenopausal women with hormone receptor-positive, human epidermal growth factor receptor 2-negative breast cancer T4 Nany or Tany N2-3
  Interventions: Drug: Tamoxifen 20mg; Drug: Anastrozole 1mg; Drug: Letrozole 2.5mg; Drug: Goserelin; Drug: Triptorelin
- postmenopausal women: postmenopausal women with hormone receptor-positive, human epidermal growth factor receptor 2-negative breast cancer T4 Nany or Tany N2-3
  Interventions: Drug: Tamoxifen 20mg; Drug: Anastrozole 1mg; Drug: Letrozole 2.5mg

INTERVENTIONS:
Drug: Tamoxifen 20mg — Selective estrogen receptor modulator
Drug: Anastrozole 1mg — Aromatase Inhibitor
Drug: Letrozole 2.5mg — Aromatase Inhibitor
Drug: Goserelin — Gonadotropin Releasing Hormone (GnRH) agonist
  Groups: premenopausal women
Drug: Triptorelin — Gonadotropin Releasing Hormone (GnRH) agonist
  Groups: premenopausal women

SUMMARY:
Neoadjuvant Endocrine Therapy for pre- and postmenopausal women with T4 Nany or TanyN2-3 estrogen receptor (ER) -positive, progrsteron receptor (PR) -positive and HER2 negative breast cancer. Real Clinical Practice in Russia.

DETAILED DESCRIPTION:
Neoadjuvant Endocrine Therapy for pre- and postmenopausal women with T4 Nany or TanyN2-3 estrogen receptor (ER) -positive, progrsteron receptor (PR) -positive and HER2 negative breast cancer. Real Clinical Practice in Russia.

Nonrandomized, retrospective clincal trial

Eligible postmenopausal women were treated with tamoxifen 20 mg, exemestane 25 mg daily, letrozole 2.5 mg daily, or anastrozole 1 mg daily before surgery

or

Eligible premenopausal women were treated with tamoxifen 20 mg, exemestane 25 mg daily, letrozole 2.5 mg daily, or anastrozole 1 mg daily in combination with ovarian suppression before surgery

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed of hormone receptor-positive (HR +), human epidermal growth factor receptor 2-negative (HER2-) invasive breast cancer T4 Nany or Tany N2-N3 premenopausal or menopausal women aged 18 years or older. No evidence of metastasis (M0) No prior hormonal, chemotherapy or radiotherapy is allowed. No breast operation other than biopsy to make diagnosis is allowed.

Postmenopausal women, defined as women meeting any of the following criteria:

Age ≥ 60 years Age ≥ 45 years with amenorrhea ≥ 12 months in the moment of breast cancer diagnosis and an intact uterus Prior bilateral ovariectomy In case previous hysterectomy, follicle stimulating hormone (FSH) and estradiol levels within the postmenopausal range (using local laboratory ranges)* * In patients previously treated with a luteinizing hormone releasing hormone (LH-RH) analogue, the last extended release formulation should have been administered more than 6 months before randomisation, and menses must not have reappeared.

For women of childbearing potential who are sexually active, agreement to use a highly effective, non-hormonal form of contraception or two effective forms of non-hormonal contraception during and for at least 6 months post-treatment.Eastern Cooperative Oncology Group (ECOG) performance status 0/1/2 No personal history of breast cancer within the last 5 years

Exclusion Criteria:

Patients non-candidate for breast surgery Patients with previously treated breast cancer during the last 5 years or receiving another concomitant anticancer treatment like chemotherapy, immunotherapy, endocrine Patient whose general clinical condition does not consider postponing surgery

Inadequate organ function, evidenced by the following laboratory results:

Absolute neutrophil count <1,500 cells/mm3 Platelet count <100,000 cells/mm3 Hemoglobin <9 g/dL Total bilirubin greater than 1,5 times the upper limit of normal (ULN) (unless the patient has documented Gilbert's syndrome) Aspartate aminotransferase (AST [SGOT]) or alanine aminotransferase (ALT [SGPT]) >2.5 x ULN Serum creatinine >2.0 mg/dL and/or 177 μmol/L clearance creatinine <50mL/min (calculated by Cockcroft-Gault method) International normalized ratio (INR) and activated partial thromboplastin time (aPTT) or partial thromboplastin time (PTT) >1.5 x ULN (unless on therapeutic coagulation) 9. Uncontrolled hypertension (systolic >150 mmHg and/or diastolic > 100 mmHg) or clinically significant (i.e. active) cardiovascular disease: cerebrovascular accident/stroke or myocardial infarction within 6 months prior to first study medication; unstable angina; CHF of New York Heart Association (NYHA) Grade II or higher; or serious cardiac arrhythmia requiring medication.

Patients with a history of long-QT syndrome or documented family history of long-QT syndrome.

QTc >470 12. serum potassium level < LLN 13. Uncontrolled intercurrent illness including but not limited to, known active infection with human immunodeficiency virus (HIV), hepatitis B or C virus or psychiatric illness/social situations that would limit compliance with study requirements.

Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Pregnant or breastfeeding patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: premenopausal or menopausal women aged 18 years or older with histologically confirmed of hormone receptor-positive (HR +), human epidermal growth factor receptor 2-negative (HER2-) invasive breast cancer T4 Nany or Tany N2-N3
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-04-15 (Actual); Primary Completion 2023-08-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
the number of patients with a Residual Cancer Burden (RCB) 0-I index as a measure of efficacy | Up to 5 years
  Residual cancer burden (RCB) is estimated from routine pathologic sections of the primary breast tumor site and the regional lymph nodes after the completion of neoadjuvant therapy. 6 variables are included in a calculation formula.

SECONDARY OUTCOMES:
clinical response in each treatment arm as defined by clinical and ultrasound examination. | Up to 5 years
Preoperative Endocrine Prognostic Index (PEPI) | Up to 5 years
  the preoperative endocrine prognostic index (PEPI)- consisting of the pathological tumor size, pathological node status, Ki67 labeling index, and ER status of residual tumors after NAE
the rates of breast conservation therapy with regard to the initially planned surgery | Up to 5 years
Disease-free survival (DFS) | Up to 5 years
  DFS event is defined as the evidence of local and/or distant recurrence, new primary breast tumour, or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Blokhin's Russian Cancer Research Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
Neoadjuvant Endocrine Therapy in Breast Cancer. Real Clinical Practice in Russia.